CLINICAL TRIAL: NCT06567431
Title: Examination of Alzheimer's Disease Biomarkers in Tears and Dry Blood Spots
Brief Title: Blood And Tears in Alzheimer's Disease
Acronym: BAT-AD
Status: Recruiting | Type: Observational
Sponsor: Danish Dementia Research Centre (Network)
Responsible Party: Sponsor
Other Study IDs: H-23078392
Record Dates: First submitted 2024-03-18; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Neurodegenerative Diseases
MeSH Terms: conditions — Neurodegenerative Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Tears and dry blood spots from fingerprick
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Alzheimer's disease: Patients diagnosed with Alzheimer's disease (AD), either MCI, mild or moderate dementia.
- Cognitive impairment due to non-Alzheimer's disease: Patients diagnosed with one of the following dementia disorders: Dementia with Lewy Bodies (DLB), Frontotemporal dementia (FTD), vascular dementia (VaD) and Normal pressure hydrocephalus (NPH).
- Controls: Patients who have undergone a diagnostic work-up in a memory clinic, but no neurodegenerative or other neurological disease was found, serve as control group.

SUMMARY:
This study aims to investigate whether biomarkers of Alzheimer's disease can be found in tearfluid, as well as dried bloodspots in patients with Alzheimer's disease, other dementia diagnoses compared to controls.

DETAILED DESCRIPTION:
Participants under investigation of a neurodegenerative disease who have a planned lumbar puncture in the Memory clinic will be invited to this study. On the same day of the lumbar puncture, tear fluid and dry blod spots will be collected.

Tear fluid is collected using Shirmer's test. Dried blood spots are obtained by a small prick in the finger with a lancet. The blood droplet is transferred onto a special piece of filter paper, where it dries.

As a sub-study, participants who have provided written consent specifically for this purpose will repeat the test with dried blood spots at home one week after participating in the study. The samples are submitted to the Memory Clinic at the participant's next scheduled appointment.

Tear fluid, dried blood spots, as well as blood and cerebrospinal fluid will be examined for AD-related pathology.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for patients:

* Lumbar puncture with CSF avaiable for analysis
* Diagnosis of Alzheimer's disease, Dementia with Lewy Bodies (DLB), Frontotemporal dementia (FTD), vascular dementia (VaD) or Normal pressure hydrocephalus (NPH)
* Of legal age.

Inclusion criteria for controls:

* Lumbar puncture with CSF avaiable for analysis
* No neurological disease.
* Of legal age.

Exclusion Criteria:

* No lumbar puncture
* Clinically assessed as unfit to participate in the project.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We aim to include 177 participants in each group. The diagnoses are based on internationally recognised diagnostic criteria for the individual diseases, and the diagnosis is made at a consensus conference by experienced specialists in the field of dementia.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
AD related biomarkers in tear fluid | Two years
  Concentrations of AD biomarkers (AB42, AB40, Ptau217, NfL, GFAP) in tear fluid in the AD-group compared to non-AD and controls.
AD related biomarkers in dry blod spots | Two years
  Concentrations of AD biomarkers (AB42, AB40, Ptau217, NfL, GFAP) in dry blot spots in the AD-group compared to non-AD and controls.

SECONDARY OUTCOMES:
Testing dry blod spots at home | Two years
  To test the feasability of dry blod spots card in a home setting - measuring concentrations of AD biomarkers in the blod cards performed at home compared to the card performed in the clinic.

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Dementia Research Centre, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No